CLINICAL TRIAL: NCT03901807
Title: A Prospective, Multicenter, Randomized, Open-Label Study to Evaluate the Efficacy and Safety of PMX Cartridge in Addition to Standard Medical Care for Patients With Endotoxemic Septic Shock
Brief Title: Safety and Efficacy of Polymyxin B Hemoperfusion (PMX) for Endotoxemic Septic Shock in a Randomized, Open-Label Study
Acronym: TIGRIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spectral Diagnostics (US) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDI-PMX-NA003
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Septic Shock; Endotoxemia
Keywords: sepsis; septic shock; severe sepsis; endotoxemia; endotoxemic; TIGRIS; PMX; Toraymyxin; EAA; Spectral Medical
MeSH Terms: conditions — Shock, Septic; Endotoxemia; Sepsis

STUDY DESIGN:
Intervention Model Description: The subjects will be randomized in a 2:1 ratio to the two groups (PMX cartridge plus standard of care: standard of care alone). A blocked randomization scheme will be used to provide approximately balanced ratio allocations to the two groups for each investigative site during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- PMX Treatment (Experimental): Standard medical care for septic shock plus treatment with the PMX cartridge (twice approximately 24 hours apart)
  Interventions: Device: Toraymyxin PMX 20R Extracorporeal Hemoperfusion Cartridge
- Control (No Intervention): Standard medical care alone

INTERVENTIONS:
Device: Toraymyxin PMX 20R Extracorporeal Hemoperfusion Cartridge — TORAYMYXIN PMX-20R (PMX) is an extracorporeal hemoperfusion cartridge intended for the selective removal of endotoxin from circulating blood through direct hemoperfusion (DHP). Each treatment will target 2 hours with a minimum of 1 ½ hours, at a flow rate of approximately 100 mL/minute, (range of 80 to 120 mL/minute).
  Arms: PMX Treatment

SUMMARY:
Prospective, multicenter, randomized, open-label study of standard of care plus the PMX cartridge versus standard of care alone in patients with endotoxemic septic shock

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, open-label trial of standard medical care plus the PMX cartridge versus standard medical care alone, in subjects with endotoxemia and septic shock. Subjects in critical care areas will be assessed for septic shock using known or suspected infection, multiple organ failure, fluid resuscitation and hypotension requiring vasopressor support as primary criteria. Subjects will meet all entry criteria for study if endotoxin activity is within the range of ≥ 0.60 to <0.90.

Eligible and consented subjects will be randomized to receive either the PMX cartridge (administered twice for 1½ to 2 hours per treatment session approximately 24 hours apart) plus standard medical care or standard medical care alone. For all randomized subjects, a follow-up visit (if they are still in the hospital) or a telephone call will be completed at Day 28 (or later) to determine their mortality status. In surviving subjects, a follow-up visit or telephone call to determine their mortality status will also take place at approximately three months (i.e. Day 90) and 12 months after the subject was randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age
2. Hypotension requiring vasopressor support: Requirement for at least one of the vasopressors listed below, at the dose shown below, for at least 2 continuous hours and no more than 30 hours

   1. Norepinephrine > 0.05mcg/kg/min
   2. Dopamine > 10 mcg/kg/min
   3. Phenylephrine > 0.4 mcg/kg/min
   4. Epinephrine > 0.05 mcg/kg/min
   5. Vasopressin > 0.03 units/min
   6. Vasopressin (any dose) in combination with another vasopressor listed above
3. The subject must have received intravenous fluid resuscitation of a minimum of 30mL/kg administered within 24 hours of eligibility
4. Documented or suspected infection defined as definitive or empiric intravenous antibiotic administration
5. The subject must have a screening multi-organ dysfunction score (MODS) >9 OR a sequential organ failure assessment (SOFA) >11, in the event a complete MODS cannot be obtained due to missing measurements
6. Endotoxin Activity Assay between ≥ 0.60 to <0.90 EA units
7. Evidence of at least 1 of the following criteria for new onset organ dysfunction that is considered to be due to the acute illness:

   1. Requirement for positive pressure ventilation via an endotracheal tube or tracheostomy tube
   2. Thrombocytopenia defined as acute onset of platelet count <150,000µ/L or a reduction of 50% from prior known levels
   3. Acute oliguria defined as urine output <0.5mL/kg/hr for at least 6 hours despite adequate fluid resuscitation

Exclusion Criteria:

1. Inability to obtain an informed consent from the subject, family member or an authorized surrogate
2. Lack of commitment for full medical support
3. Inability to achieve or maintain a minimum mean arterial pressure (MAP) of ≥ 65mmHg despite vasopressor therapy and fluid resuscitation
4. Subject has end-stage renal disease and requires chronic dialysis
5. There is clinical support for non-septic shock such as:

   1. Acute pulmonary embolus
   2. Transfusion reaction
   3. Severe congestive heart failure (e.g. NYHA Class IV, ejection fraction < 35%)
6. Subject has had chest compressions as part of CPR during this hospitalization without immediate return to communicative state
7. Subject has had an acute myocardial infarction (AMI) within the past 4 weeks
8. Subject has uncontrolled hemorrhage (acute blood loss requiring > 3 UPC in the past 24 hours)
9. Major trauma within 36 hours of screening
10. Subject has severe granulocytopenia (leukocyte count less than 500 cells/mm3) or severe thrombocytopenia (platelet count less than 30,000 cells/mm3)
11. HIV infection in association with a last known or suspected CD4 count of <50/mm3
12. Subject's baseline state is non-communicative
13. Subject has sustained extensive third-degree burns within the past 7 days
14. Body weight < 35 kg (77 pounds)
15. Known hypersensitivity to Polymyxin B
16. Subject has known sensitivity or allergy to heparin or has a history of heparin associated thrombocytopenia (H.I.T.)
17. Subject is currently enrolled in an investigational drug or device trial
18. Subject has been previously enrolled in the current trial
19. Any other condition, that in the opinion of the investigator, would preclude the subject from being a suitable candidate for enrollment, such as end-stage chronic illness (eg. lack of source control and bowel necrosis) with no reasonable expectation of survival to hospital discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Day 28 mortality comparison | 28 days
  The primary objective is to compare the safety and efficacy of the PMX cartridge (Toraymyxin) based on mortality at 28 days in patients with septic shock and endotoxemia who are treated with standard medical care plus the use of the PMX cartridge, versus patients who receive standard medical care alone.

SECONDARY OUTCOMES:
Day 90 mortality comparison | 90 days
  compare mortality at 90 days post baseline in each group
MAP comparison | 3 days
  compare changes in mean arterial blood pressure (MAP) from Day 0 to Day 3 in each group
Vasopressor dose comparison | 3 days
  compare the changes in vasopressor doses from Day 0 to Day 3 in each group
Survival time comparison | 28 days
  compare the survival time from baseline to death within 28 days in each group
Day 28 mortality comparison for patients on norepinephrine >0.1 mcg/kg/min | 28 days
  compare mortality at 28 days post baseline for patients with baseline norepinephrine dose >0.1 mcg/kg/min in each group
Day 14 mortality comparison | 14 days
  compare mortality at 14 days post baseline in each group
Vasopressor use comparison | 3 days
  compare total duration of vasopressor use from Day 0 to Day 3 in each group
12 month mortality comparison | 12 months
  compare mortality at 12 months post baseline in each group

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California, San Francisco, San Francisco, California
  - Pulmonary Associates, Boulder, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Louisiana State University Health Shreveport, Shreveport, Louisiana
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Cooper Health System, Camden, New Jersey
  - Rutgers, The State University of New Jersey, Piscataway, New Jersey
  - Mt Sinai Hospital, New York, New York
  - Stony Brook University, Stony Brook, New York
  - UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CHI Memorial, Chattanooga, Tennessee
  - Parkridge Hospital, Chattanooga, Tennessee
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Institute for Extracorporeal Life Support, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
There are no plans for sharing IPD at this time.

REFERENCES:
- [Derived] Bellomo R, Mehta RL, Forni LG, Zarbock A, Ostermann M, Ronco C; Acute Disease Quality Initiative Hemoadsorption Working Group. Hemoadsorption. Clin J Am Soc Nephrol. 2024 Jan 12;19(6):803-806. doi: 10.2215/CJN.0000000000000433. Epub 2024 Jan 12. No abstract available. PMID 38214917